CLINICAL TRIAL: NCT07081867
Title: Comparison of Postoperative Analgesic Efficacy of Preoperatively Performed Sacral Erector Spinae Plane Block and Supra-Inguinal Fascia Iliaca Block in Patients Undergoing Surgery for Hip Fracture
Brief Title: Comparison of Sacral Erector Spinae Plane Block and Supra-Inguinal Fascia Iliaca Block for Analgesia After Hip Fracture Surgery
Status: Completed | Type: Observational
Sponsor: Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization (Other)
Responsible Party: Principal Investigator, Beyzanur Aydoğdu, Resident Doctor, Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Other Study IDs: CT-ERHO-AR-BA-01
Record Dates: First submitted 2025-07-09; First posted 2025-07-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Hip Fracture Surgery; Postoperative Pain Management; Regional Anesthesia; Elderly Patients
Keywords: Nerve Block; Anesthesia, Regional; Hip Fractures; Postoperative Pain; Analgesia; Visual Analog Scale; Pain Measurement
MeSH Terms: conditions — Hip Fractures; Pain, Postoperative; Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SIFIB Group: Patients who underwent Supra-Inguinal Fascia Iliaca Block (n=40)
  Interventions: Procedure: Supra-inguinal Fascia Iliaca Block (SIFIB)
- SESPB Group: Patients who underwent Sacral Erector Spinae Plane Block (n=37)
  Interventions: Procedure: Sacral Erector Spinae Plane Block (SESPB)

INTERVENTIONS:
Procedure: Supra-inguinal Fascia Iliaca Block (SIFIB) — Ultrasound-guided injection of 40 mL of 0.25% bupivacaine between the iliacus muscle and fascia iliaca via a supra-inguinal approach, performed preoperatively for postoperative analgesia in patients undergoing hip fracture surgery under spinal anesthesia.
  Groups: SIFIB Group
Procedure: Sacral Erector Spinae Plane Block (SESPB) — Ultrasound-guided injection of 40 mL of 0.25% bupivacaine into the fascial plane deep to the erector spinae muscle at the sacral level (S2), performed preoperatively for postoperative analgesia in patients undergoing hip fracture surgery under spinal anesthesia.
  Groups: SESPB Group

SUMMARY:
This study compares the postoperative analgesic effectiveness of Sacral Erector Spinae Plane Block (SESPB) and Supra-Inguinal Fascia Iliaca Block (SIFIB) in patients undergoing hip fracture surgery. Both techniques are regional anesthesia methods aiming to reduce postoperative pain and opioid consumption. The study evaluates pain scores, opioid requirements, mobilization times, and hospital discharge times to determine which block provides more effective pain management in different postoperative periods.

DETAILED DESCRIPTION:
Hip fractures are common injuries among elderly patients, often resulting in high rates of morbidity and mortality. Effective postoperative pain management plays a critical role in reducing complications such as delayed mobilization, deep vein thrombosis, pneumonia, and prolonged hospitalization.

Regional anesthesia techniques, including Sacral Erector Spinae Plane Block (SESPB) and Supra-Inguinal Fascia Iliaca Block (SIFIB), have gained popularity as part of multimodal analgesia strategies that aim to minimize opioid use and improve postoperative comfort. However, there is limited evidence comparing these two techniques directly.

In this prospective observational study, patients aged 65 and older undergoing hip fracture surgery under spinal anesthesia were included. After obtaining informed consent, patients received either SESPB or SIFIB for postoperative analgesia in addition to the standard anesthetic protocol.

Pain levels were assessed using the Visual Analog Scale (VAS) at 1, 6, 12, and 24 hours after surgery. Additional data such as total opioid consumption within 24 hours, time to first analgesic requirement, mobilization time, and length of hospital stay were recorded.

The results demonstrated that patients who received SIFIB had significantly lower pain scores in the early postoperative period (1st hour), while patients who received SESPB experienced better pain relief in the late postoperative period (24th hour). No significant differences were observed between the groups in terms of total opioid consumption, mobilization time, or hospital stay duration. No complications related to the block procedures were reported.

This study suggests that both SESPB and SIFIB are safe and effective regional anesthesia techniques for postoperative pain management in hip fracture surgeries. The selection between these blocks may be based on the desired onset and duration of analgesia, with SIFIB providing superior early pain control and SESPB offering more prolonged analgesic effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 65 years and older
* Patients undergoing surgery for hip fractures under spinal anesthesia
* Patients who are oriented and cooperative
* Patients who have signed an informed consent form

Exclusion Criteria:

* Patients with contraindications for spinal anesthesia
* Patients with Alzheimer's disease or dementia, and those who are non-oriented or non-cooperative
* Patients with major organ failure (such as heart, liver, or kidney failure)
* Patients who decline to participate in the study
* Patients classified as American Society of Anesthesiologists (ASA) Physical Status IV or higher
* Patients with pathological fractures or bone metastasis

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients aged 65 years and older who underwent hip fracture surgery under spinal anesthesia at Prof. Dr. Cemil Taşçıoğlu City Hospital between January and June 2025. Only patients who provided written informed consent and met the inclusion criteria were enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
Postoperative Pain Scores | At 1 hour, 6 hours, 12 hours, and 24 hours postoperatively.
  Pain intensity measured using the Visual Analog Scale (VAS), ranging from 0 to 10, where 0 indicates no pain and 10 indicates the worst pain imaginable. Pain scores will be recorded at specific postoperative time points: 1st, 6th, 12th, and 24th hours.
Time to First Postoperative Analgesic Requirement | Up to 48 hours postoperatively.
  Time interval from end of surgery to the first request for analgesia.
Total Postoperative Opioid Consumption | A week
  The total amount of opioids required by patients during the postoperative period.
Time to First Mobilization | From the end of surgery until first mobilization, typically within 24 to 48 hours postoperatively
  The time until patients' first mobilization (walking or standing) after surgery.

SECONDARY OUTCOMES:
Length of Hospital Stay | Up to 14 days postoperatively.
  Duration from the day of surgery to the day of hospital discharge, measured in calendar days.
Block-Related Complications | A week
  Possible complications following Sacral Erector Spinae Plane Block (SESPB) and Supra-Inguinal Fascia Iliaca Block (SIFIB), such as nerve injury, infection, hematoma, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Beyzanur Aydogdu, Principal Investigator — Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization
Locations (1):
- Prof. Dr. Cemil Tascıoglu Education and Research Hospital Organization, Istanbul, Sisli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual patient data will not be shared due to patient privacy requirements and ethical board restrictions.